CLINICAL TRIAL: NCT02013284
Title: Is Our Microbiome a Predictor of Cardiac Risk?
Brief Title: Is Our Microbiome a Predictor of Cardiac Risk
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amir Lerman, Amir Lerman, MD, Mayo Clinic
Other Study IDs: 13-007084
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (50 cc) and stool samples will be collected on consenting participants. Participants will have the option of allowing us to store samples for future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to determine a relationship between a person's flora/bacteria in their gut (the intestinal microbiome) and their risk of cardiovascular disease. Investigators will look at inflammatory markers in the blood and also look at the genome of the bacteria in the gut.

DETAILED DESCRIPTION:
Investigators will look at inflammatory markers in the blood and also look at the genome of the bacteria in the gut. This research is being done because Investigators believe that there is a connection between the way food is digested by a person's gut bacteria and the development of atherosclerosis (hardening of the arteries) and cardiovascular disease. The ultimate goal of this research is to eventually determine if changes to the gut bacteria can prevent cardiovascular disease or disease progression.

ELIGIBILITY:
Inclusion Criteria:

Anyone undergoing cardiac catheterization for suspected coronary artery disease over age 18.

Exclusion Criteria:

1. Patients currently on long-term antibiotics who cannot stop them for at least 2 weeks prior to providing a stool sample.
2. Patients on chronic laxatives who cannot stop for at least 2 weeks prior to stool collection.
3. Patients on probiotics and cannot stop for 2 weeks prior to giving a stool sample (yogurt is ok).
4. Patients who are unable to provide a stool sample to Mayo Clinic within 24 hours of collection utilizing Fed Ex overnight mail (i.e. people overseas who are unable to provide a sample before leaving the USA.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consenting participants who are undergoing coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2013-11; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
50 cc blood obtained during angiogram and used for Endothelial Progenitor Cells analysis using antibodies for inflammatory markers. Plasma collection will be done for antibody analysis. Buffy coats will be frozen and stored for future genetic analysis. | Blood samples will be obtained during the diagnostic angiogram.

SECONDARY OUTCOMES:
Stool samples will be collected to compare the fecal microbiota of patients with mild, moderate and severe coronary artery disease. | Two weeks after the angiogram

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No